CLINICAL TRIAL: NCT04655092
Title: Extension Study of P1101 in Japanese Patients Who Have Completed Phase 2 Single Arm Study in Polycythemia Vera (PV) Patients (Study A19-201) or Phase 3 Study in Essential Thrombocythemia (ET) Patients (Study P1101 ET)
Brief Title: Extension Study of P1101 After Completion of Phase 2 Study in PV Patients or Phase 3 Study in ET Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A20-201
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Polycythemia Vera (PV)
Keywords: Myeloproliferative Neoplasms
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders

STUDY DESIGN:
Intervention Model Description: Conventional treatment based on phlebotomies, low-dose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of P1101 (ropeginterferon alfa-2b) once every 2 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P1101 (Ropeginterferon alfa-2b) (Experimental): Conventional treatment based on phlebotomies, lowdose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of pegylated prolineinterferon alpha-2b (P1101, Ropeginterferon alfa-2b) once every 2 weeks.
  Interventions: Biological: P1101 (Ropeginterferon alfa-2b)

INTERVENTIONS:
Biological: P1101 (Ropeginterferon alfa-2b) — The subjects who have completed the 52-week treatment duration in Study A19-201 will be treated with P1101, starting at the dose at Week 50. The dose during this study may be increased or decreased up to 500 μg depending on the condition. This study will be continued as a post-marketing clinical study after acquisition of the marketing approval of P1101.

SUMMARY:
This is a Phase 3 open-label, multicenter, single arm study designed to evaluate the efficacy and safety and tolerability of P1101 patient with PV or ET in long-term.

DETAILED DESCRIPTION:
The study is to evaluate the long-term safety and efficacy of P1101 in PV or ET patients who participated in Study A19-201 or Study P1101 ET. The subjects who have completed the 52-week P1101 treatment duration in Study A19-201 will start treatment with P1101 at the dose at Week 50. The subjects who have completed the follow-up/end-of-study visit in Study P1101 ET will start treatment with P1101 at the dose at Week 50. The subjects who were treated with anagrelide will start treatment with P1101 at a dose of 250 μg. The dose of P1101 during this study may be increased or decreased up to 500 μg depending on the condition.

Evaluation of safety will include assessing vital signs, clinical safety laboratory tests, physical examinations, ECG evaluation, heart ECHO, lung X-ray, ECOG performance status, ocular examination, and AEs.

Efficacy evaluations, safety assessments, and immunogenicity evaluations of P1101 will be performed.

Evaluation of efficacy will include clinical laboratory assessments, allelic burden measurements of CALR, JAK-2, and MPL, spleen size measurements, bone marrow sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the 52-week treatment duration in Study A19-201 and are considered by the investigator or sub investigator to be eligible for participation in this study
* Patients who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients who are considered by the investigator or sub investigator to be ineligible for continued treatment with P1101

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maintenance rate of phlebotomy-free complete hematologic response (CHR) every 52 weeks | Through study completion, an average of 2 year
  CHR will be defined as follows.
  * Hematocrit <45% phlebotomy-free (absence of phlebotomy during the previous 12 weeks)
  * Platelet count ≤ 400 x 10^9/L
  * WBC count ≤ 10 x 10^9/L

SECONDARY OUTCOMES:
Changes in hematocrit every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Changes in white blood cell every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Changes in platelet count every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Changes in red blood cell count every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Changes in spleen size every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Necessity of phlebotomy | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Proportion of subjects without thrombotic or hemorrhagic events | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201
Changes in JAK2 V617F mutant allelic burden value every 52 weeks over time | Through study completion, an average of 2 year
  Baseline is defined as Week 52 in Study A19-201

OTHER OUTCOMES:
Bone marrow histological remission (optional) | Through study completion, an average of 2 year
  Bone marrow histological remission was defined as the disappearance of hypercellularity and trilineage growth (panmyelosis), and absence of >grade 1 reticulin fibrosis in the subjects who gave informed consent in Study A19-201

CONTACTS AND LOCATIONS:
Overall Officials: Keita Kirito, MD, Principal Investigator — University of Yamanashi Hospital
Locations (6):
- Japan (6):
  - Ehime University Hospital, Toon-shi, Ehime
  - Mie University Hospital, Tsu, Mie-ken
  - Osaka University Hospital, Suita-shi, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: No